CLINICAL TRIAL: NCT03752528
Title: Evaluation of Long-term Buprenorphine Plasma Exposure in Subjects Who Received at Least 2 Subcutaneous (SC) Injections of Extended-release Buprenorphine (SUBLOCADE™) in Phase III Studies
Brief Title: Evaluation of Long-term Buprenorphine Plasma Exposure
Status: Completed | Type: Observational
Sponsor: Indivior Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: INDV-6000-402
Record Dates: First submitted 2018-11-21; First posted 2018-11-26 (Actual); Results first posted 2020-08-03 (Actual); Last update posted 2020-08-21 (Actual); Status verified 2020-08

CONDITIONS: Opioid-use Disorder
MeSH Terms: conditions — Opioid-Related Disorders

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — PK plasma samples to assess buprenorphine concentrations
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Part A Cohort: Representative data set of participants from study RB-US-13-0003 or both studies RB-US-13-0003 and INDV-6000-301 who received at least 2 doses of SUBLOCADE 12-36 months prior. Part A consists of a single visit (Visit 1) for both screening and collection of blood and urine samples.
  Interventions: Diagnostic Test: Blood sample collection; Diagnostic Test: Urine sample collection
- Part B Cohort: Part A participants with a quantifiable (i.e. positive) result for buprenorphine and/or norbuprenorphine and a non-quantifiable (i.e. negative) result for naloxone continue in the study for two additional visits (Visits 2 and 3) which are conducted approximately 30 days apart during which blood and urine samples are collected.
  Interventions: Diagnostic Test: Blood sample collection; Diagnostic Test: Urine sample collection

INTERVENTIONS:
Diagnostic Test: Blood sample collection — Determination of buprenorphine and norbuprenorphine plasma concentrations
Diagnostic Test: Urine sample collection — Urine sample for determination of free buprenorphine and free norbuprenorphine concentrations, qualitative UDS for opioids, quantitative UDS for buprenorphine, norbuprenorphine and naloxone, and determination of creatinine concentration

SUMMARY:
The study objective is to characterise the long-term plasma exposure to buprenorphine after stopping SUBLOCADE treatment. There are no interventions planned.

This multicentre investigation will enroll participants from Study RB-US-13-0003 (NCT02510014) or both Studies RB-US-13-0003 and INDV-6000-301 (NCT02896296) and who received at least 2 subcutaneous (SC) injections of SUBLOCADE.

There are two parts to the study:

Part A consists of a single visit during which urine samples are collected to measure free buprenorphine and free norbuprenorphine concentrations; qualitative urine drug samples (UDS) for opioids, including buprenorphine; quantitative UDS for buprenorphine, norbuprenorphine and naloxone; and determination of creatinine concentration. Blood samples are collected for the determination of buprenorphine and norbuprenorphine plasma concentrations.

Results on the quantitative UDS performed in Part A determine enrollment in Part B: participants who provide a quantifiable (i.e., positive) result for buprenorphine and/or norbuprenorphine and a non-quantifiable (i.e., negative) result for naloxone meet continuation criteria to move on to Part B if Part B is still open to enrolment. Part B consists of two visits 30 days apart in which the same tests are run as were done in Part A.

DETAILED DESCRIPTION:
Data indicate that after discontinuing SUBLOCADE patients may have detectable concentrations of buprenorphine in plasma and urine for 12 months or longer. Previous Phase II/III studies did not evaluate the pharmacokinetics (PK) of buprenorphine beyond 2 months after the last injection; this study will characterize the long-term plasma exposure starting at least 12 months after the last injection. The study will also assess relationships between plasma drug concentrations, free drug concentrations in urine and urine drug screen (UDS) results in order to provide refined guidance to patients and physicians with respect to long-term exposure to buprenorphine after stopping SUBLOCADE treatment.

ELIGIBILITY:
Inclusion Criteria:

* Participated in Study RB-US-13-0003 or both Studies RB-US-13-0003 and INDV-6000-301 and received at least 2 subcutaneous (SC) injections of SUBLOCADE
* Within 12 to 36 months post his or her last SUBLOCADE injection at the time of the Screening Visit
* Female individuals of childbearing potential must agree to have a pregnancy test administered prior to enrollment and throughout the study. Pregnancy does not prohibit participation
* Willing to adhere to study procedures and provide written informed consent prior to the start of any study procedures.

Exclusion Criteria:

* Received SUBLOCADE or any other long-acting buprenorphine product at any time after ending their participation in Study RB-US-13-0003 or Study INDV-6000-301
* Taken any buprenorphine (prescribed or illicit) within 3 weeks prior to the Screening visit (study Part A, Visit 1)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Subjects who participated in either of the studies listed above and who received their last SUBLOCADE injection within 12 to 30 months of the Screening visit. A maximum of 30 subjects may continue to Part B and will return for 2 additional visits 30 days apart.
Sampling Method: Non-Probability Sample
Enrollment: 53 (Actual)
Dates: Start 2019-02-19 (Actual); Primary Completion 2019-07-18 (Actual); Study Completion 2019-07-18 (Actual)

CONTACTS AND LOCATIONS:
Locations (11):
- United States (11):
  - Pathway Healthcare, Hamilton, Alabama
  - Meridian Research, Tampa, Florida
  - Phoenix Medical Research, Prairie Village, Kansas
  - Adams Clinical, Watertown, Massachusetts
  - Hassman Research Institute, Berlin, New Jersey
  - Neurobehavioral Clinical Research, North Canton, Ohio
  - Pahl Research, Oklahoma City, Oklahoma
  - SP Research, Oklahoma City, Oklahoma
  - CODA, Portland, Oregon
  - Clinical Research Associates of Central PA, LLC, Altoona, Pennsylvania
  - Pillar Research, Richardson, Texas

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: All investigators sites were in the U.S.
Pre-assignment Details: 54 subjects were screened. One did not meet eligibility criteria.
Groups:
- All Study Participants: All study participants who enrolled into the Part A Cohort. These participants previously participated in study RB-US-13-0003 or both studies RB-US-13-0003 and INDV-6000-301 and who received at least 2 doses of SUBLOCADE 12-36 months prior. Some of the participants continued into study Part B after completing Part A.
Period: Part A
Arm/Group | All Study Participants
Started | 53
Completed | 51
Not Completed | 2
Not completed — Lost to Follow-up | 1
Not completed — Protocol Violation | 1
Period: Part B
Arm/Group | All Study Participants
Started (Requirement: positive for buprenorphine and/or norbuprenorphine and negative for naloxone in Part A) | 24
Completed | 20
Not Completed | 4
Not completed — Protocol Violation | 1
Not completed — Study terminated by sponsor | 3

BASELINE CHARACTERISTICS:
Population: Safety Analysis Set
Arm/Group | All Study Participants
Number analyzed (Participants) | 53
Age, Continuous [Mean (Standard Deviation); unit: years] | 43.0 (11.46)
Age, Customized [Count of Participants; unit: Participants]
  18 - 44 years | 32
  45 - 64 years | 19
  .>= 65 years | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21
  Male | 32
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3
  Not Hispanic or Latino | 50
  Unknown or Not Reported | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Black or African American | 16
  White | 37
Region of Enrollment [Number; unit: participants]
  United States | 53
Weight [Mean (Standard Deviation); unit: kg] | 79.7 (18.51)
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] | 26.5 (5.58)
Body Mass Index Group [Count of Participants; unit: Participants]
  < 18.5 kg/m^2 | 1
  >= 18.5 and < 25 kg/m^2 | 24
  >= 25 and < 30 kg/m^2 | 15
  >= 30 kg/m^2 | 13

OUTCOME MEASURES:

1. Primary Outcome: Qualitative Urinary Drug Screen (UDS) for Buprenorphine in Parts A + B
Description: The qualitative UDS (immunoassay) is the primary test used for the initial screening for opioids in patients in clinical practice. It provides only a qualitative assessment of buprenorphine exposure (i.e., positive or negative) with a low limit of quantification (LLOQ) of 5 ng/mL. The qualitative UDS is reported for Part A Cohort (Visit 1) and Part B Cohort (Visits 1, 2 and 3).
  Participants' last subcutaneous injections of extended release buprenorphine (SUBLOCADE™) was 22 - 38 months prior during previous phase III studies.
Time Frame: Days 1, 30, 60
Population: Full analysis set includes participants who have at least one measure of buprenorphine or norbuprenorphine concentration in plasma or in urine in Part A. Four participants who tested positive for naloxone in urine were excluded from summary results. One participant was terminated from the study prior to Part B, Visit 2.
Measure: Count of Participants; unit: Participants
Groups:
- Part A Cohort: Visit 1: Representative data set of participants from study RB-US-13-0003 or both studies RB-US-13-0003 and INDV-6000-301 who received at least 2 doses of SUBLOCADE 12-36 months prior. Part A consists of a single visit (Visit 1) for both screening and collection of blood and urine samples.
- Part B Cohort: Visit 1: Part A participants with a quantifiable (i.e. positive) result for buprenorphine and/or norbuprenorphine and a non-quantifiable (i.e. negative) result for naloxone continue in the study for two additional visits (Part B, Visits 2 and 3). This cohort reports Visit 1 results for those participants who continued into Part B of the study.
- Part B Cohort: Visit 2: Part A participants with a quantifiable (i.e. positive) result for buprenorphine and/or norbuprenorphine and a non-quantifiable (i.e. negative) result for naloxone continue in the study for two additional visits (Part B, Visits 2 and 3). This cohort reports Visit 2 (Day 30) results for those participants who continued into Part B of the study.
- Part B Cohort: Visit 3: Part A participants with a quantifiable (i.e. positive) result for buprenorphine and/or norbuprenorphine and a non-quantifiable (i.e. negative) result for naloxone continue in the study for two additional visits (Part B, Visits 2 and 3). This cohort reports Visit 3 (Day 60) results for those participants who continued into Part B of the study.
Arm/Group | Part A Cohort: Visit 1 | Part B Cohort: Visit 1 | Part B Cohort: Visit 2 | Part B Cohort: Visit 3
Number analyzed (Participants) | 49 | 24 | 23 | 20
Participants
  Positive | 27 | 19 | 16 | 15
  Negative | 22 | 5 | 7 | 5

2. Primary Outcome: Quantitative Urine Drug Screen (UDS) for Buprenorphine and Norbuprenorphine in Parts A + B
Description: The quantitative UDS measures both buprenorphine and its glucuronide, or both norbuprenorphine and its glucuronide, with an LLOQ of 2 ng/mL. It is typically used by physicians for the confirmation of a positive result on the qualitative UDS.
  Data are reported for Part A Cohort (Visit 1) and Part B Cohort (Visits 1, 2 and 3).
  For Bup+Nor (abbreviation for Buprenorphine + Norbuprenorphine), the result is negative if results for both are negative, the result is positive if either result is positive. If both are missing/not available, or one is negative and the other is missing/not evaluable, the result is "Not Available"
  Participants' last subcutaneous injections of extended release buprenorphine (SUBLOCADE™) was 22 - 38 months prior during previous phase III studies.
Time Frame: Days 1, 30, 60
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Part A Cohort: Visit 1 | Part B Cohort: Visit 1 | Part B Cohort: Visit 2 | Part B Cohort: Visit 3
Number analyzed (Participants) | 49 | 24 | 23 | 20
Participants
  Buprenorphine - Positive | 31 | 23 | 19 | 17
  Buprenorphine - Negative | 18 | 1 | 4 | 3
  Buprenorphine - Not Available | 0 | 0 | 0 | 0
  Norbuprenorphine - Positive | 29 | 21 | 19 | 17
  Norbuprenorphine - Negative | 19 | 2 | 4 | 3
  Norbuprenorphine- Not Available | 1 | 1 | 0 | 0
  Bup + Nor - Positive | 32 | 24 | 20 | 18
  Bup + Nor - Negative | 17 | 0 | 3 | 2
  Bup + Nor - Not Available | 0 | 0 | 0 | 0

3. Primary Outcome: Urine Free Drug Test for Buprenorphine and Norbuprenorphine in Parts A + B
Description: The urine free drug test only measures the "free" buprenorphine and "free" norbuprenorphine (without their glucuronides) with an LLOQ of 0.02 ng/mL.
  Data are reported for Part A Cohort (Visit 1) and Part B Cohort (Visits 1, 2 and 3).
  For Bup+Nor (abbreviation for Buprenorphine + Norbuprenorphine), the result is negative if results for both are negative, the result is positive if either result is positive. If both are missing/not available, or one is negative and the other is missing/not evaluable, the result is "Not Available"
  Participants' last subcutaneous injections of extended release buprenorphine (SUBLOCADE™) was 22 - 38 months prior during previous phase III studies.
Time Frame: Days 1, 30, 60
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Part A Cohort: Visit 1 | Part B Cohort: Visit 1 | Part B Cohort: Visit 2 | Part B Cohort: Visit 3
Number analyzed (Participants) | 49 | 24 | 23 | 20
Participants
  Buprenorphine - Positive | 30 | 19 | 17 | 17
  Buprenorphine - Negative | 19 | 5 | 5 | 3
  Buprenorphine - Not Available | 0 | 0 | 1 | 0
  Norbuprenorphine - Positive | 46 | 24 | 21 | 20
  Norbuprenorphine - Negative | 3 | 0 | 1 | 0
  Norbuprenorphine- Not Available | 0 | 0 | 1 | 0
  Bup + Nor - Positive | 46 | 24 | 21 | 20
  Bup + Nor - Negative | 3 | 0 | 1 | 0
  Bup + Nor - Not Available | 0 | 0 | 1 | 0

4. Primary Outcome: Plasma Drug Test for Buprenorphine and Norbuprenorphine in Parts A + B
Description: A sensitive liquid chromatography with tandem mass spectrometry (LC-MS/MS) method was used to assess the plasma exposure to buprenorphine and norbuprenorphine, its major metabolite. The LLOQ was 0.02 ng/mL for both analytes, which is much lower than the LLOQ of plasma/serum assays conducted by diagnostic laboratories.
  Data are reported for Part A Cohort (Visit 1) and Part B Cohort (Visits 1, 2 and 3).
  For Bup+Nor (abbreviation for Buprenorphine + Norbuprenorphine), the result is negative if results for both are negative, the result is positive if either result is positive. If both are missing/not available, or one is negative and the other is missing/not evaluable, the result is "Not Available"
  Participants' last subcutaneous injections of extended release buprenorphine (SUBLOCADE™) was 22 - 38 months prior during previous phase III studies.
Time Frame: Days 1, 30, 60
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Part A Cohort: Visit 1 | Part B Cohort: Visit 1 | Part B Cohort: Visit 2 | Part B Cohort: Visit 3
Number analyzed (Participants) | 49 | 24 | 23 | 20
Participants
  Buprenorphine - Positive | 32 | 20 | 18 | 16
  Buprenorphine - Negative | 15 | 3 | 4 | 3
  Buprenorphine - Not Available | 2 | 1 | 1 | 1
  Norbuprenorphine - Positive | 20 | 12 | 11 | 11
  Norbuprenorphine - Negative | 27 | 11 | 11 | 8
  Norbuprenorphine- Not Available | 2 | 1 | 1 | 1
  Bup + Nor - Positive | 32 | 20 | 18 | 16
  Bup + Nor - Negative | 15 | 3 | 4 | 3
  Bup + Nor - Not Available | 2 | 1 | 1 | 1

ADVERSE EVENTS:
Time Frame: Day 1 to Day 60
Description: Only adverse events (AEs) associated with study assessments and/or study conduct were collected.
  Since there is no study drug for this study, no treatment emergent AE is defined for this study.
Arm/Group | All Study Participants
All-Cause Mortality (participants affected / at risk) | 0/53
Serious Adverse Events (participants affected / at risk) | 0/53
Other Adverse Events (participants affected / at risk) | 0/53

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Proposed publications shall be submitted to Sponsor 30 days prior to submission for publication, and may be withheld for an additional period, up to 90 days, to allow Sponsor to file patent applications. If a multi-center publication isn't submitted for publication within 12 months of the conclusion of the Study at all sites, or is published in a shorter period, the results from the institution's site may be published individually.

DOCUMENTS (2):
  • Study Protocol (2019-04-22): https://cdn.clinicaltrials.gov/large-docs/28/NCT03752528/Prot_000.pdf
  • Statistical Analysis Plan (2019-05-22): https://cdn.clinicaltrials.gov/large-docs/28/NCT03752528/SAP_001.pdf